CLINICAL TRIAL: NCT01882283
Title: Effects of Black Tea Intake on Serum Lipids in Mildly Hypercholesterolemic Adults A Randomized Diet-controlled Crossover Trial
Brief Title: Effects of Black Tea Intake on Serum Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 10205345-A2; M01RR000400 (NIH)
Record Dates: First submitted 2013-06-17; First posted 2013-06-20 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Hypercholesterolemia
Keywords: serum lipids; cholesterol; serum cholesterol; black tea; flavonoids; crossover trial; randomized control trial; diet controlled
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tea Treatment Group (Experimental): 5 cups brewed tea beverage per day for 28 days, brewed from 700 mg of black tea solids per cup
  Interventions: Dietary Supplement: Tea Treatment Group
- Placebo Group (Placebo Comparator): 5 cups tea-like placebo per day for 28 days. Placebo was exactly matched to tea except for flavonoid composition. Placebo was flavonoid-free.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Tea Treatment Group — This intervention was a crossover trial, during which each patient experienced both placebo and tea treatment arms
  Other Names: Brewed black tea beverage
  Arms: Tea Treatment Group
Dietary Supplement: Placebo
  Arms: Placebo Group

SUMMARY:
A diet-controlled clinical trial which attempts to provide estimates of the effect of black tea consumption on serum lipids under tightly controlled conditions, including a controlled diet. Mildly hypercholesterolemic individuals (total cholesterol levels between 4.9 and 6.7 mmol/L, 190 and 260 mg/dl), non-smoking, chronic disease-free individuals were enrolled in a 15-week, double blind, randomized crossover trial, during which they consumed a controlled low-flavonoid diet plus 5 cups of black tea or a tea-like placebo over two 4-week treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* between 45-65 years old
* mildly hypercholesterolemic (total cholesterol levels between 4.9 and 6.7 mmol/L, 190 and 260 mg/dl)
* high-density lipoprotein cholesterol (HDL-C) between 0.9 and 1.6 mmol/L (35 and 65 mg/dl)
* triglyceride (TG) concentrations below 6.8 mmol/L (600 mg/dl)
* habitually consumed a typical American diet with low dietary flavonoid intake (<4 one-half cup servings of fruits and vegetables/day) and low intake (<1 serving/day) of soy-rich foods, nuts, herbs, and spices (besides salt and pepper)
* aspartate aminotransferase (AST) between 0 and 55 mg/L
* creatinine between 70.7 and 150.3 mmol/L (0.8 and 1.7 mg/dl)
* glucose between 3.3 and 6.4 mmol/L (60 and 115 mg/dl)

Exclusion Criteria:

* current smoker
* usage of high amounts of antioxidant vitamin supplements (>3 times the Recommended Dietary Allowance (RDA) of vitamins E, C, and selenium, or >10 mg/day of beta carotene)
* had been diagnosed with diabetes, coagulation disorders, chronic pulmonary disease, current active malignancy, renal disease requiring dialysis, malabsorption, or gastrointestinal disorders, or had a history of cardiovascular disease.
* antihypertensive, immunosuppressive, cholesterol lowering, or anticoagulant medications
* consuming >3 servings of alcohol daily
* Pre-menopausal (women)

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2002-04; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Serum lipid levels | 4 weeks
  Serum lipid levels (total cholesterol, LDL-C, HDL-C, triglycerides, LDL-C+HDL-C fraction, LDL-C/HDL-C ratio) were assessed at the end of a 28-day treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Myron Gross, PhD, Principal Investigator — University of Minnesota
Locations (1):
- General Clinical Research Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Troup R, Hayes JH, Raatz SK, Thyagarajan B, Khaliq W, Jacobs DR Jr, Key NS, Morawski BM, Kaiser D, Bank AJ, Gross M. Effect of black tea intake on blood cholesterol concentrations in individuals with mild hypercholesterolemia: a diet-controlled randomized trial. J Acad Nutr Diet. 2015 Feb;115(2):264-271.e2. doi: 10.1016/j.jand.2014.07.021. Epub 2014 Sep 27. PMID 25266246